CLINICAL TRIAL: NCT02662660
Title: Postoperative Pain After Laparoscopic Sleeve Gastrectomy: Comparison of Isolated Intravenous Analgesia, Epidural Analgesia Associated With Analgesia iv and Port-sites Infiltration With Bupivacaine Associated With Analgesia iv
Brief Title: Analgesia iv vs Epidural Analgesia vs Port-sites Infiltration After Laparoscopic Sleeve Gastrectomy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital General Universitario Elche (Other)
Responsible Party: Principal Investigator, Jaime Ruiz-Tovar, MD, PhD, MD, PhD, Hospital General Universitario Elche
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HGUE 16-03
Record Dates: First submitted 2016-01-17; First posted 2016-01-25 (Estimated); Last update posted 2016-01-25 (Estimated); Status verified 2016-01

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine; Analgesia, Epidural; Dipyrone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Port-sites infiltration:Bupivacaine0,25% (Experimental): Port-sites infiltration will be performed with 10 ml of Bupivacaine 0.25%, applying 2 ml under the aponeurotic layer in each port. Associated intravenous analgesia will include Metamizole 2g/8h and Acetaminophen 1g/8h, alternating every 4 hours.
  Interventions: Drug: Port-sites infiltration:Bupivacaine0.25%; Drug: Metamizole and Acetaminophen iv
- Epidural analgesia:Levobupivacaine0.125% (Experimental): Epidural analgesia consists in the placement of a thoracic epidural catheter inserted at the level T6-T7 and administration of a continuous perfusion of Levobupivacaine 0.125% 6ml/h.
  Associated intravenous analgesia will include Metamizole 2g/8h and Acetaminophen 1g/8h, alternating every 4 hours.
  Interventions: Drug: Epidural analgesia:Levobupivacaine0,125%; Drug: Metamizole and Acetaminophen iv
- Metamizole and Acetaminophen iv (Active Comparator): Associated intravenous analgesia will include Metamizole 2g/8h and Acetaminophen 1g/8h, alternating every 4 hours.
  Interventions: Drug: Metamizole and Acetaminophen iv

INTERVENTIONS:
Drug: Port-sites infiltration:Bupivacaine0.25% — Port-sites infiltration will be performed with 10 ml of Bupivacaine 0.25%, applying 2 ml under the aponeurotic layer in each port.
  Other Names: Port-sites infiltration with bupivacaine
  Arms: Port-sites infiltration:Bupivacaine0,25%
Drug: Epidural analgesia:Levobupivacaine0,125% — Port-sites infiltration will be performed with 10 ml of Bupivacaine 0.25%, applying 2 ml under the aponeurotic layer in each port.
  Other Names: Epidural analgesia
  Arms: Epidural analgesia:Levobupivacaine0.125%
Drug: Metamizole and Acetaminophen iv — Associated Intravenous analgesia include Metamizole 2g/8h and Acetaminophen 1g/8h, alternating every 4 hours.
  Other Names: Analgesia iv

SUMMARY:
A prospective randomized study of patients undergoing laparoscopic sleeve gastrectomy between 2012 and 2015 will be performed. Patients will be divided into 3 groups: Analgesia iv exclusively (Group 1), epidural analgesia+analgesia iv (Group 2) and port-sites infiltration+analgesia iv (Group 3). Pain will be quantified by means of a Visual Analogic Scale and morphine rescue needs were determined 24 hours after surgery.

DETAILED DESCRIPTION:
A prospective randomized study of patients undergoing laparoscopic sleeve gastrectomy between 2012 and 2015 will be performed. Patients will be randomized using a computerized simple randomization scheme in a 1:1:1 ratio into 3 groups: those patients receiving only intravenous analgesia (Group 1), those ones receiving intravenous analgesia associated to epidural analgesia (Group 2) and those patients receiving intravenous analgesia associated with port-sites infiltration with bupivacaine. Pain quantification as measured by Visual Analogic Scale (VAS), ranging from 0 (absence of pain) to 10 (unbearable pain) will be evaluated 24 hours after surgery.

ELIGIBILITY:
Inclusion Criteria:

* body mass index (BMI) >40 Kg/m2
* BMI > 35 Kg/m2 with the presence of comorbidities associated to obesity

Exclusion Criteria:

* patients undergoing other bariatric techniques
* severe underlying cardiovascular diseases
* chronic renal failure
* hepatic dysfunction
* previous foregut surgery
* patients with any contraindication for bariatric surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2012-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Postoperative pain measured by Visual Analogic Scale | 24 hours after surgery
  Postoperative pain will be measured by Visual Analogic Scale (VAS), ranging from 0 (absence of pain) to 10 (unbearable pain) 24 hours after surgery,

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Duran, MD, PhD, Study Director — Hospital General Elche

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ruiz-Tovar J, Munoz JL, Gonzalez J, Zubiaga L, Garcia A, Jimenez M, Ferrigni C, Duran M. Postoperative pain after laparoscopic sleeve gastrectomy: comparison of three analgesic schemes (isolated intravenous analgesia, epidural analgesia associated with intravenous analgesia and port-sites infiltration with bupivacaine associated with intravenous analgesia). Surg Endosc. 2017 Jan;31(1):231-236. doi: 10.1007/s00464-016-4961-3. Epub 2016 May 13. PMID 27177956